CLINICAL TRIAL: NCT00046228
Title: A Muticenter, Randomized, Double-blind, Placebo Controlled Trial Comparing the Efficacy and Safety of Reteplease and Abciximab Combination Therapy With Abciximab Alone Administered Early or Just Prior to Primary Primary Percutaneous Coronary Intervention for Acute Myocardial Infarction.
Brief Title: A Study of Abciximab and Reteplase When Administered Prior to Catherization After a Myocardial Infarction (Finesse)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR005410; FINESSE; CR005410
Record Dates: First submitted 2002-09-24; First posted 2002-09-25 (Estimated); Results first posted 2009-05-15 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; percutaneous coronary intervention; abciximab; reteplase; safety and efficacy
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab; reteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): Abciximab; reteplase; abciximab placebo; abciximab 0.25 mg/kg bolus; 1-2, 5 unit boluses; placebo bolus; 0.125 ¼g/kg/min, max 10 ¼g/min infusion x 12h
  Interventions: Drug: abciximab placebo; reteplase placebo, abciximab, abciximab; Drug: Abciximab; reteplase; abciximab placebo; abciximab
- 002 (Experimental): abciximab; reteplase placebo; abciximab placebo; abciximab 0.25 mg/kg bolus; 1-2 placebo boluses; placebo bolus; 0.125 ¼g/kg/min, max 10 ¼g/min infusion x 12h
  Interventions: Drug: Abciximab; reteplase; abciximab placebo; abciximab; Drug: abciximab; reteplase placebo; abciximab placebo; abciximab
- 003 (Experimental): abciximab placebo; reteplase placebo, abciximab, abciximab placebo bolus; 1-2 placebo bolus; 0.25 mg/kg bolus; 0.125 ¼g/kg/min, max 10 ¼g/min infusion x 12h
  Interventions: Drug: abciximab; reteplase placebo; abciximab placebo; abciximab; Drug: abciximab placebo; reteplase placebo, abciximab, abciximab

INTERVENTIONS:
Drug: abciximab placebo; reteplase placebo, abciximab, abciximab — placebo bolus; 1-2 placebo bolus; 0.25 mg/kg bolus; 0.125 ¼g/kg/min, max 10 ¼g/min infusion x 12h
  Arms: 001
Drug: Abciximab; reteplase; abciximab placebo; abciximab — 0.25 mg/kg bolus; 1-2, 5 unit boluses; placebo bolus; 0.125 ¼g/kg/min, max 10 ¼g/min infusion x 12h
  Arms: 002
Drug: abciximab; reteplase placebo; abciximab placebo; abciximab — 0.25 mg/kg bolus; 1-2 placebo boluses; placebo bolus; 0.125 ¼g/kg/min, max 10 ¼g/min infusion x 12h
  Arms: 003
Drug: abciximab placebo; reteplase placebo, abciximab, abciximab — placebo bolus; 1-2 placebo bolus; 0.25 mg/kg bolus; 0.125 ¿g/kg/min, max 10 ¿g/min infusion x 12h
  Arms: 003
Drug: abciximab; reteplase placebo; abciximab placebo; abciximab — 0.25 mg/kg bolus; 1-2 placebo boluses; placebo bolus; 0.125 ¿g/kg/min, max 10 ¿g/min infusion x 12h
  Arms: 002
Drug: Abciximab; reteplase; abciximab placebo; abciximab — 0.25 mg/kg bolus; 1-2, 5 unit boluses; placebo bolus; 0.125 ¿g/kg/min, max 10 ¿g/min infusion x 12h
  Arms: 001

SUMMARY:
The purpose of this study is to determine whether abciximab given in combination with reteplase, before patients have a coronary intervention (a standard treatment where a catheter is inserted into the heart artery to get blood flowing past the clot), is safe and effective in the treatment of heart attacks compared to only abciximab given during coronary intervention.

DETAILED DESCRIPTION:
The purpose of this medical research study is to determine whether abciximab given in combination with reteplase, before patients have a coronary intervention (a standard treatment where a catheter is inserted into the heart artery to get blood flowing past the clot), is safe and effective in the treatment of heart attacks compared to only abciximab given during coronary intervention. This medical research study will also help determine if the combination of abciximab and reduced dose reteplase will decrease the risk of death, and reduce complications of a heart attack at 90 days compared to abciximab alone which is a standard treatment.

Patients will receive either abciximab and reteplease or abciximab alone. Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive either abciximab and reteplease or abciximab and placebo into a vein in their arm for up to 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have prolonged, continuous (lasting at least 20 minutes) signs and symptoms of A heart attack not eliminated with nitrates and onset within 6 hours of randomization,and confirmation by Electrocardiogram

Exclusion Criteria:

* Low risk clinical presentation
* patients who will not be undergoing a catherization within 4 hours of the qualifying Electrocardiogram

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2461 (Actual)
Dates: Start 2002-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (227):
- United States (52):
  - Phoenix, Arizona
  - Covina, California
  - Modesto, California
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Weston, Florida
  - Harvey, Illinois
  - Rock Island, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Lewiston, Maine
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Pontiac, Michigan
  - St Louis, Missouri
  - Brooklyn, New York
  - Flushing, New York
  - Mineola, New York
  - New York, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Westlake, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - Sellersville, Pennsylvania
  - Upland, Pennsylvania
  - Wormleysburg, Pennsylvania
  - York, Pennsylvania
  - Pawtucket, Rhode Island
  - Providence, Rhode Island
  - Spartanburg, South Carolina
  - Bristol, Tennessee
  - Kingsport, Tennessee
  - Amarillo, Texas
  - Galveston, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Bremerton, Washington
  - Marshfield, Wisconsin
  - Waukesha, Wisconsin
- Argentina (6):
  - Adrogué
  - Buenos Aires
  - Corrientes
  - Merlo
  - Rosario
  - San Martín
- Austria (5):
  - Bruck an der Mur
  - Deutschlandsberg
  - Innsbruck
  - Linz
  - Vienna
- Belgium (10):
  - Antwerp
  - Bonheiden
  - Eeklo
  - Ghent
  - Herentals
  - Mechelen
  - Reet
  - Turnhout
  - Waregem
  - Westmalle
- Bulgaria (4):
  - Dimitrovgrad
  - Haskovo
  - Plovdiv
  - Sofia
- Canada (3):
  - Edmonton, Alberta
  - Montreal, Quebec
  - Repentigny, Quebec
- Czechia (41):
  - Benesov U Prahy
  - Bílovec
  - Boskovice
  - Brno
  - Bruntál
  - Čáslav
  - České Budějovice
  - Český Krumlov
  - Havíøov 1
  - Hodonín
  - Hradec Králové
  - Hranice
  - Jeseník
  - Jičín
  - Jihlava
  - Karniva-Ray N/A
  - Kyjov
  - Most
  - Nový Jičín
  - Odry
  - Olomouc
  - Ostrava
  - Písek
  - Poruba
  - Prague
  - Praha 10 N/A
  - Prostějov
  - Přerov
  - Strakonice
  - Svitavy
  - Šumperk
  - Tábor
  - Teplice
  - Trutnov
  - Tøebíè 1
  - Tøinec 1
  - Ústí nad Labem
  - Ústí nad Orlicí
  - Valašské Meziříčí
  - Vyškov
  - Znojmo
- Denmark (13):
  - Esbjerg
  - Frederikshavn
  - Hjÿrring N/A
  - Horsens
  - Kÿbenhavn Nv N/A
  - Kÿbenhavn Sud N/A
  - Kÿbenhavn Ÿ
  - Odense
  - Randers
  - Silkeborg
  - Viborg
  - Ÿlborg
  - Ÿrhus N
- France (8):
  - Besançon
  - Colmar
  - Metz
  - Nancy
  - Nancy Cedex N/A
  - Nîmes
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (18):
  - Aachen
  - Bad Nauheim
  - Bad Segeberg
  - Bremen
  - Dresden
  - Eschweiler
  - Friedberg
  - Fulda
  - Hamburg
  - Kaltenkirchen
  - Magdeburg
  - Mannheim
  - Meißen
  - München
  - Münster
  - Pfaffenhofen
  - Radebeul
  - Schönebeck
- Israel (2):
  - Jerusalem
  - Ramat Gan
- Leeuwarden, Netherlands
- Poland (33):
  - Będzin
  - Bielsko-Biala
  - Bolesławiec
  - Brzeg
  - Częstochowa
  - Gdansk
  - Gdynia Poland
  - Gliwice
  - Gmina Końskie
  - Gorlice
  - Grójec
  - Jastrzębie Zdrój
  - Katowice
  - Konin
  - Kościerzyna
  - Krakow
  - Lodz
  - Nowy Dwor M
  - Nysa
  - Opole
  - Piotrkow Trybunalski
  - Poznan
  - Radomsko
  - Ruda Śląska
  - Skierniewice
  - Swidnica
  - Tychy
  - Ustroń
  - Warsaw
  - Warszawa Poland
  - Wroclaw
  - Zabrze
  - Żyrardów
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Târgu Mureş
- South Africa (3):
  - Arcadia Pretoria N/A
  - Cape Town Western Province
  - Roodepoort Central Gauteng
- Spain (5):
  - Alicante
  - Barcelona
  - Madrid
  - Santander
  - Santiago de Compostela
- Gothenburg, Sweden
- Switzerland (3):
  - Basel
  - Bruderholz
  - Liestal
- United Kingdom (15):
  - Antrim
  - Belfast
  - Brighton
  - Chichester
  - Durham
  - Glasgow
  - London
  - Manchester
  - Middlesbrough
  - Plymouth
  - Portadown
  - Saint Leonards-on-Sea
  - Southampton
  - Stockton-on-Tees
  - Worthing

REFERENCES:
- [Result] Ellis SG, Armstrong P, Betriu A, Brodie B, Herrmann H, Montalescot G, Neumann FJ, Smith JJ, Topol E; Facilitated Intervention with Enhanced Reperfusion Speed to Stop Events Investigators. Facilitated percutaneous coronary intervention versus primary percutaneous coronary intervention: design and rationale of the Facilitated Intervention with Enhanced Reperfusion Speed to Stop Events (FINESSE) trial. Am Heart J. 2004 Apr;147(4):E16. doi: 10.1016/j.ahj.2003.07.025. PMID 15077099
- [Result] Ellis SG, Tendera M, de Belder MA, van Boven AJ, Widimsky P, Janssens L, Andersen HR, Betriu A, Savonitto S, Adamus J, Peruga JZ, Kosmider M, Katz O, Neunteufl T, Jorgova J, Dorobantu M, Grinfeld L, Armstrong P, Brodie BR, Herrmann HC, Montalescot G, Neumann FJ, Effron MB, Barnathan ES, Topol EJ; FINESSE Investigators. Facilitated PCI in patients with ST-elevation myocardial infarction. N Engl J Med. 2008 May 22;358(21):2205-17. doi: 10.1056/NEJMoa0706816. PMID 18499565
- [Derived] Montalescot G, Ellis SG, de Belder MA, Janssens L, Katz O, Pluta W, Ecollan P, Tendera M, van Boven AJ, Widimsky P, Andersen HR, Betriu A, Armstrong P, Brodie BR, Herrmann HC, Neumann FJ, Effron MB, Lu J, Barnathan ES, Topol EJ; Facilitated INtervention with Enhanced Reperfusion Speed to Stop Events Investigators. Enoxaparin in primary and facilitated percutaneous coronary intervention A formal prospective nonrandomized substudy of the FINESSE trial (Facilitated INtervention with Enhanced Reperfusion Speed to Stop Events). JACC Cardiovasc Interv. 2010 Feb;3(2):203-12. doi: 10.1016/j.jcin.2009.11.012. PMID 20170878
- [Derived] Herrmann HC, Lu J, Brodie BR, Armstrong PW, Montalescot G, Betriu A, Neuman FJ, Effron MB, Barnathan ES, Topol EJ, Ellis SG; FINESSE Investigators. Benefit of facilitated percutaneous coronary intervention in high-risk ST-segment elevation myocardial infarction patients presenting to nonpercutaneous coronary intervention hospitals. JACC Cardiovasc Interv. 2009 Oct;2(10):917-24. doi: 10.1016/j.jcin.2009.06.018. PMID 19850249
- [Derived] Ellis SG, Tendera M, de Belder MA, van Boven AJ, Widimsky P, Andersen HR, Betriu A, Savonitto S, Adamus J, Peruga JZ, Hamankiewicz M, Pluta W, Oldroyd K, Ecollan P, Janssens L, Armstrong P, Brodie BR, Herrmann HC, Montalescot G, Neumann FJ, Effron MB, Barnathan ES, Topol EJ; FINESSE Investigators. 1-year survival in a randomized trial of facilitated reperfusion: results from the FINESSE (Facilitated Intervention with Enhanced Reperfusion Speed to Stop Events) trial. JACC Cardiovasc Interv. 2009 Oct;2(10):909-16. doi: 10.1016/j.jcin.2009.07.009. PMID 19850248
- See also: A Study of Abciximab and Reteplase When Administered Prior to Catheterization After a Myocardial Infarction - Finesse — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=15&filename=CR005410_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 20 countries. The FINESSE (Facilitated INtervention with Enhanced Reperfusion Speed to Stop Events) study began enrollment in August 2002. It was planned that approximately 3,000 subjects would be enrolled. Because of enrollment difficulty, subject enrollment was stopped on 30 Dec 2006.
Pre-assignment Details: A total of 2,461 subjects were enrolled in the study according to the sponsor's clinical trial management system. Out of 2461 subjects, 2,452 subjects were randomly assigned to the 3 treatment groups.
Groups:
- Primary PCI Group: Abciximab (bolus + 12 hr infusion) initiated just prior to primary percutaneous coronary intervention (PCI)
- Abciximab Facilitated PCI Group: Abciximab (bolus) administered as soon as possible after randomization, 12 hour infusion initiated prior to PCI
- Reteplase/Abciximab Facilitated PCI Group: Abciximab (bolus) + reteplase (5 U + 5 U double bolus for subjects < 75 years of age; 5 U single bolus for subjects ≥ 75 years of age), abciximab 12 hour infusion initiated prior to PCI
Period: 90 Days
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Started | 806 | 818 | 828
Completed | 793 (The number completed includes subjects who died or were seen for a visit within specified window.) | 810 (The number completed includes subjects who died or were seen for a visit within specified window.) | 813 (The number completed includes subjects who died or were seen for a visit within specified window.)
Not Completed | 13 | 8 | 15
Period: 1 Year
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Started | 806 (This is the number of participants that were originally randomized to the trial.) | 818 (This is the number of participants that were originally randomized to the trial.) | 828 (This is the number of participants that were originally randomized to the trial.)
Completed | 787 (The number completed includes subjects who died or were seen for a visit within specified window.) | 804 (The number completed includes subjects who died or were seen for a visit within specified window.) | 816 (The number completed includes subjects who died or were seen for a visit within specified window)
Not Completed | 19 | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group | Total
Number analyzed (Participants) | 806 | 818 | 828 | 2452
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.4) | 61.9 (11.8) | 62.6 (11.4) | 62.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 216 | 219 | 642
  Male | 599 | 602 | 609 | 1810

OUTCOME MEASURES:

1. Primary Outcome: The Composite of All-Cause Mortality or Complications of MI at 90 Days.
Description: Occurs within 90 days and is composite of all-cause mortality or complications of myocardial infarction (MI) (rehospitalization or emergency department visit for congestive heart failure (CHF), cardiogenic shock, or resuscitated ventricular fibrillation occurring > 48 hours after randomization).
Time Frame: 90 days
Population: Population is the intent-to-treat subjects. The intent-to-treat population is defined as all subjects randomly assigned to a treatment group and classified according to the randomization assignment.
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 806 | 818 | 828
participants | 86 | 86 | 81
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the primary PCI in terms of the primary efficacy outcome. Assuming the relative risk reduction for the reteplase/abciximab facilitated PCI group versus the Primary PCI group is 15% in lower risk, 25% in medium risk, and 35% in high risk, the power of this comparison (1,000 subjects per group) is 83.4 %; Test type: Superiority or Other; p = 0.551, Log Rank — The null hypothesis was tested at the significance level of 0.049. If it is significant, the significance level of null hypotheses tested in the analyses 2 and 3 will be adjusted according to the modified Hochberg approach; Independent Clinical Endpoints Committee confirmed components of primary endpoint except for death & resuscitated v fib assessed by the investigator); Hazard Ratio (HR) = 0.91, 95% CI [0.67 to 1.23]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; The null hypothesis is if abciximab facilitated PCI is the same as the primary PCI in terms of the primary efficacy outcome. Assuming the relative risk reduction for the Abciximab facilitated PCI versus the Primary PCI group is 12.7%, in lower risk, 17.9% in medium risk, and 25.0% in high risk, the power of this comparison (1000 subjects per group) is 54.1%; Test type: Superiority or Other; p = 0.858, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI [0.72 to 1.31]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the abciximab facilitated PCI in terms of the primary efficacy outcome. Assuming the relative risk reduction for the reteplase/abciximab facilitated PCI versus the abciximab facilitated PCI group is 2.6% in lower risk, 8.7% in medium risk, and 13.3% in high risk, the power of this comparison (1,000 subjects per group) is 13.5%; Test type: Superiority or Other; p = 0.676, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI [0.69 to 1.27]

2. Secondary Outcome: Complications of MI as Defined in the Primary Outcome Measure Through 90 Days
Description: The complications of myocardial infarction (MI) is defined as any event of rehospitalization or emergency department visit for CHF, cardiogenic shock, or resuscitated ventricular fibrillation occurring > 48 hours after randomization.
Time Frame: 90 Days
Population: Population is the intent-to-treat subjects. The intent-to-treat population is defined as all subjects that have been randomly assigned to a treatment group and classified according to the randomization assignment.
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 806 | 818 | 828
participants | 72 | 61 | 61
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the primary PCI in complications of MI within 90 days; Test type: Superiority or Other; p = 0.247, Chi-squared; Odds Ratio (OR) = 0.81, 95% CI [0.57 to 1.16]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; The null hypothesis is if abciximab facilitated PCI is the same as the primary PCI in complications of MI within 90 days; Test type: Superiority or Other; p = 0.278, Chi-squared; Odds Ratio (OR) = 0.82, 95% CI [0.58 to 1.17]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the abciximab facilitated PCI in complications of MI within 90 days; Test type: Superiority or Other; p = 0.944, Chi-squared; Odds Ratio (OR) = 0.99, 95% CI [0.68 to 1.43]

3. Secondary Outcome: All-Cause Mortality Through 90 Days
Description: All cause mortality occurred through 90 days from randomization.
Time Frame: 90 days
Population: Population is the intent-to-treat subjects. The intent-to-treat population is defined as all randomized subjects classified according to the randomization assignment.
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 806 | 818 | 828
participants | 36 | 45 | 43
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if retaplase/abciximab facilitated PCI is the same as the primary PCI in 90-day all cause mortality; Test type: Superiority or Other; p = 0.494, Chi-squared; Odds Ratio (OR) = 1.17, 95% CI [0.74 to 1.84]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; The null hypothesis is if abciximab facilitated PCI is the same as the primary PCI in 90-day all cause mortality; Test type: Superiority or Other; p = 0.338, Chi-squared; Odds Ratio (OR) = 1.25, 95% CI [0.79 to 1.95]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if retaplase/abciximab facilitated PCI is the same as the abciximab facilitated PCI in 90-day all cause mortality; Test type: Superiority or Other; p = 0.781, Chi-squared; Odds Ratio (OR) = 0.94, 95% CI [0.61 to 1.45]

4. Secondary Outcome: Subjects With ST-Segment Resolution > 70% From Baseline at 60 to 90 Minutes Following Randomization
Time Frame: 60 to 90 minutes
Population: Population is the intent-to-treat subjects who were selected for evaluation by electrocardiogram (ECG) core laboratory.Subjects, who were not evaluable for a 60-90 minute ECG, were considered not having a ST segment resolution.
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 405 | 432 | 424
participants | 75 | 85 | 108
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if retaplase/abciximab facilitated PCI is the same as the primary PCI in ST-segment resolution >70% from baseline; Test type: Superiority or Other; p = 0.016, Chi-squared; Odds Ratio (OR) = 1.50, 95% CI [1.08 to 2.10]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; The null hypothesis is if abciximab facilitated PCI is the same as the primary PCI in ST-segment resolution >70% from baseline; Test type: Superiority or Other; p = 0.670, Chi-squared; Odds Ratio (OR) = 1.08, 95% CI [0.76 to 1.52]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if retaplase/abciximab facilitated PCI is the same as the abciximab facilitated PCI in ST-segment resolution >70% from baseline; Test type: Superiority or Other; p = 0.042, Chi-squared; Odds Ratio (OR) = 1.40, 95% CI [1.01 to 1.93]

5. Secondary Outcome: All-Cause Mortality Through 1 Year
Description: All-cause mortality through 1 year from randomization.
Time Frame: 1 year
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 806 | 818 | 828
participants | 56 | 60 | 52
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.603, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI [0.62 to 1.32]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.765, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI [0.73 to 1.52]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.415, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI [0.59 to 1.24]

6. Other Pre Specified Outcome: Subjects With Intracranial Hemorrhage (Including Hemorrhagic Transformation) Through Discharge/Day 7
Description: All cases of cerebrovascular event were confirmed by a CEC (Clinical Endpoints Committee).
Time Frame: Discharge/Day 7
Population: The population was defined as all subjects who were randomized and treated with any study agent, including those who discontinued for any reasons. Subjects randomized and treated was classified according to the study drug(s) received.
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 795 | 805 | 814
participants | 1 | 0 | 5
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the primary PCI in the risk of ICH; Test type: Superiority or Other; p = 0.218, Fisher Exact
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; The null hypothesis is if abciximab facilitated PCI is the same as the primary PCI in the risk of ICH; Test type: Superiority or Other; p = 0.497, Fisher Exact
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the abciximab facilitated PCI in the risk of ICH; Test type: Superiority or Other; p = 0.062, Fisher Exact

7. Other Pre Specified Outcome: Subjects With Non Intracranial Thrombolysis In Myocardial Infarction (TIMI) Bleeding Events Through Discharge/Day 7
Description: Subjects with nonintracranial TIMI bleeding (either major or minor) through discharge/day 7, originating from vascular instrumentation sites, non-instrument related bleeding, as well as overall, were examined.
Time Frame: Discharge/Day 7
Population: as for outcome 6
Measure: Number; unit: participant
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 795 | 805 | 814
participant | 55 | 81 | 118
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the primary PCI in the risk of non-ICH TIMI bleeding events; Test type: Superiority or Other; p < 0.001, Fisher Exact; Odds Ratio (OR) = 2.28, 95% CI [1.63 to 3.19]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; The null hypothesis is if abciximab facilitated PCI is the same as the primary PCI in the risk of non-ICH TIMI bleeding events; Test type: Superiority or Other; p = 0.025, Fisher Exact; Odds Ratio (OR) = 1.51, 95% CI [1.05 to 2.15]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; The null hypothesis is if reteplase/abciximab facilitated PCI is the same as the abciximab facilitated PCI in the risk of non-ICH TIMI bleeding events; Test type: Superiority or Other; p = 0.008, Fisher Exact; Odds Ratio (OR) = 1.52, 95% CI [1.12 to 2.05]

8. Other Pre Specified Outcome: Subjects With Severe Thrombocytopenia Through Discharge/Day 7
Description: Severe thrombocytopenia is defined as platelet count < 50,000 cells/μL.
Time Frame: Discharge/Day 7
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 795 | 805 | 814
participants | 11 | 16 | 16
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.439, Fisher Exact
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.438, Fisher Exact
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 1.000, Fisher Exact

9. Other Pre Specified Outcome: Subjects With Any Investigator Reported Bleeding Events Through Discharge/Day 7
Time Frame: Discharge/Day 7
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 795 | 805 | 814
participants | 139 | 178 | 271
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.020, Fisher Exact
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p < 0.001, Fisher Exact

10. Other Pre Specified Outcome: Subjects With Pre-Specified Complications of Index Myocardial Infarction Through Discharge/Day 7
Description: Number of subjects with one or more of the following: 2nd or 3rd Degree AVB, Asystole, Sustained V Tach, A Fib/Flutter, EMD/Pulseless Electrical Activity, Heart Failure, Tamponade, Myocardial Rupture, Papillary Muscle Rupture, Ventricular Septal Defect, Pulmonary Embolism, Systemic Arterial Embolism and/or Pericarditis/Pericardial Effusion.
Time Frame: Discharge/Day 7
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Number analyzed (Participants) | 806 | 818 | 828
participants | 128 | 122 | 120
Statistical Analysis 1: Comparison: Primary PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.434, Chi-squared; Odds Ratio (OR) = 0.90, 95% CI [0.69 to 1.18]
Statistical Analysis 2: Comparison: Primary PCI Group vs Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.589, Chi-squared; Odds Ratio (OR) = 0.93, 95% CI [0.71 to 1.22]
Statistical Analysis 3: Comparison: Abciximab Facilitated PCI Group vs Reteplase/Abciximab Facilitated PCI Group; Test type: Superiority or Other; p = 0.809, Chi-squared; Odds Ratio (OR) = 0.97, 95% CI [0.74 to 1.27]

ADVERSE EVENTS:
Arm/Group | Primary PCI Group | Abciximab Facilitated PCI Group | Reteplase/Abciximab Facilitated PCI Group
Serious Adverse Events (participants affected / at risk) | 159/795 | 182/805 | 175/814
Other Adverse Events (participants affected / at risk) | 0/795 | 0/805 | 0/814
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary PCI Group (N=795) | Abciximab Facilitated PCI Group (N=805) | Reteplase/Abciximab Facilitated PCI Group (N=814)
Coronary stenosis (Cardiac disorders) | 23 | 38 | 27
Shock cardiogenic (Cardiac disorders) | 4 | 9 | 13
Unstable angina (Cardiac disorders) | 4 | 2 | 6
Myocardial infarction (Cardiac disorders) | 6 | 10 | 5
Angina pectoris (Cardiac disorders) | 2 | 3 | 4
Congestive heart failure (Cardiac disorders) | 0 | 3 | 4
Myocardial ischemia (Cardiac disorders) | 1 | 1 | 4
Cardiac failure (Cardiac disorders) | 3 | 5 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 3 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 2
Chronic congestive heart failure (Cardiac disorders) | 0 | 0 | 1
Heart disorder (Cardiac disorders) | 0 | 0 | 1
Myocardial rupture (Cardiac disorders) | 2 | 2 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Spiral coronary artery dissection (Cardiac disorders) | 0 | 0 | 1
Stable angina pectoris (Cardiac disorders) | 0 | 0 | 1
Tricuspid insufficiency (Cardiac disorders) | 0 | 0 | 1
Anginal pain (Cardiac disorders) | 1 | 0 | 0
Aortic stenosis (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 2 | 0
Coronary artery perforation (Cardiac disorders) | 0 | 2 | 0
Coronary in-stent restenosis (Cardiac disorders) | 0 | 1 | 0
Coronary restenosis (Cardiac disorders) | 1 | 0 | 0
Endocarditis (Cardiac disorders) | 1 | 0 | 0
Left ventricular ejection fraction decreased (Cardiac disorders) | 1 | 0 | 0
Mitral insufficiency (Cardiac disorders) | 2 | 0 | 0
Mitral regurgitation (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Ventricular septal defect (Cardiac disorders) | 0 | 1 | 0
Fibrillation ventricular (Cardiac disorders) | 26 | 21 | 16
Cardiac arrest (Cardiac disorders) | 5 | 2 | 3
Tachycardia ventricular (Cardiac disorders) | 2 | 5 | 2
AV block complete (Cardiac disorders) | 0 | 0 | 1
AV block third degree (Cardiac disorders) | 1 | 1 | 1
Junctional bradycardia (Cardiac disorders) | 0 | 0 | 1
Nonsustained ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Arrhythmia ventricular (Cardiac disorders) | 0 | 1 | 0
Asystolia (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 2 | 0
Atrial fibrillation paroxysmal (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
AV block second degree (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrhythmia nos (Cardiac disorders) | 0 | 1 | 0
Cardiac rhythm disturbance (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary arrest (Cardiac disorders) | 1 | 0 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 1 | 0
Intraventricular conduction defect (Cardiac disorders) | 1 | 0 | 0
Tachycardia atrial paroxysmal (Cardiac disorders) | 1 | 0 | 0
Ventricular bigeminy (Cardiac disorders) | 1 | 0 | 0
Ventricular febrillation paroxysm (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 7
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Breathing difficult (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleuritis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Repiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory tract lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Breathlessness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural exudate (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia interstitial (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atherosclerosis (Cardiac disorders) | 14 | 4 | 14
Hypotension (Cardiac disorders) | 1 | 0 | 2
Syncope (Cardiac disorders) | 1 | 2 | 2
Blood pressure high (Cardiac disorders) | 0 | 0 | 1
Hypertension (Cardiac disorders) | 2 | 0 | 1
Transient hypotension (Cardiac disorders) | 0 | 0 | 1
Collapse (Cardiac disorders) | 1 | 1 | 0
Hypertension arterial (Cardiac disorders) | 1 | 0 | 0
Hypovolemic shock (Cardiac disorders) | 1 | 0 | 0
Septic shock (Cardiac disorders) | 0 | 1 | 0
Shock (Cardiac disorders) | 1 | 0 | 0
Chest pain (General disorders) | 10 | 19 | 12
Death (General disorders) | 0 | 2 | 1
Non-anginal pain (General disorders) | 0 | 0 | 1
Non-ischemic chest pain (General disorders) | 0 | 1 | 1
Allergic reaction (General disorders) | 1 | 0 | 0
Allergic reaction to diagnostic agent (General disorders) | 1 | 0 | 0
Incarcerated abdonimal hernia (General disorders) | 1 | 0 | 0
Inguinal hernia (General disorders) | 0 | 1 | 0
Interstitial fluid increased (General disorders) | 0 | 1 | 0
Intolerance induced (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Musculoskeletal pain (General disorders) | 0 | 1 | 0
Nontoxic drug overdose (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Esophageal reflux (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Polyp (Gastrointestinal disorders) | 0 | 0 | 1
Nontropical sprue (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Preploric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Digestion impaired (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric pain (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
Stomach upset (Gastrointestinal disorders) | 0 | 1 | 0
Acute renal failure (Renal and urinary disorders) | 2 | 1 | 4
Urinary tract infection (Renal and urinary disorders) | 1 | 2 | 2
Chronic renal failure (Renal and urinary disorders) | 0 | 0 | 1
Creatinine increased (Renal and urinary disorders) | 0 | 0 | 1
Renal function decreased (Renal and urinary disorders) | 0 | 0 | 1
Urethral disorder nos (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Acute renal insufficiency (Renal and urinary disorders) | 0 | 1 | 0
Bladder stricture (Renal and urinary disorders) | 0 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Pyelonephritis (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 0
Renal insufficiency (Renal and urinary disorders) | 0 | 2 | 0
Hemorrhagic stroke (Vascular disorders) | 0 | 0 | 2
Gastric hemorrhage (Vascular disorders) | 0 | 0 | 1
GI hemorrhage (Vascular disorders) | 2 | 1 | 1
GI hemorrhage - upper (Vascular disorders) | 1 | 0 | 1
Hematoma (Vascular disorders) | 1 | 1 | 1
Hemoptysis (Vascular disorders) | 1 | 0 | 1
Hemorrhage nos (Vascular disorders) | 0 | 1 | 1
Hematemesis (Vascular disorders) | 2 | 0 | 0
Hemorrhage rectum (Vascular disorders) | 0 | 1 | 0
Pulmonary hemorrhage (Vascular disorders) | 1 | 0 | 0
Puncture site hematoma (Vascular disorders) | 0 | 1 | 0
Retroperitoneal hemorrhage (type unknown) (Vascular disorders) | 1 | 0 | 0
Vomiting blood (Vascular disorders) | 1 | 0 | 0
Stroke (Vascular disorders) | 3 | 2 | 3
Claudication intermittent (Vascular disorders) | 0 | 0 | 2
Arterial stenosis (Vascular disorders) | 1 | 0 | 1
Pseudoaneurysm (Vascular disorders) | 0 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 1
Cerebral infarction (Vascular disorders) | 0 | 1 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 3 | 0
Claudication (Vascular disorders) | 1 | 0 | 0
Extracardiact arterial aneurysm (Vascular disorders) | 1 | 0 | 0
Peripheral ischemia (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Transient ischemic attack (Vascular disorders) | 1 | 0 | 0
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pulmonary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pulmonary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma nos (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cyst malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thrombosis coronary artery (Vascular disorders) | 1 | 0 | 2
Thrombosis cardiac chamber (Vascular disorders) | 0 | 0 | 1
Atheroembolism limb (Vascular disorders) | 0 | 1 | 0
Embolism pulmonary (Vascular disorders) | 2 | 3 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis venous deep (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis leg (Vascular disorders) | 1 | 0 | 0
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Skeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Adult onset diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Fever (Infections and infestations) | 0 | 0 | 1
Infection bacterial (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 2 | 0
Wound healing impaired (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 2 | 1 | 0
Epilepsy grand mal (Nervous system disorders) | 0 | 0 | 1
Pre-syncope (Nervous system disorders) | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Gall bladder distention (Hepatobiliary disorders) | 0 | 0 | 1
Hepatobiliary dysfunction (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Anemia microcytic (Blood and lymphatic system disorders) | 0 | 1 | 0
Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Delirium tremens (Psychiatric disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 1 | 1
Ventricular aneurysm (Cardiac disorders) | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 2 | 0
Breath shortness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Left ventricular thrombus (Vascular disorders) | 2 | 2 | 2
Phlebothrombosis (Vascular disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1
Anemia iron deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0
Renal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Some AEs were collected separately per protocol and are reported as "Other Pre-Specified Outcomes Measures".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days